CLINICAL TRIAL: NCT03485339
Title: Substance Misuse To Psychosis for Ketamine (SToP-K) -Who is At Risk? A Case-Control Study in Ketamine and Non-Ketamine-Using Substance Abusers
Brief Title: Substance Misuse To Psychosis for Ketamine (SToP-K)
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: SToP-K_CC
Record Dates: First submitted 2018-03-19; First posted 2018-04-02 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Ketamine Abuse; Psychotic Disorders; Substance Use Disorders; Schizophrenia; Genetic Predisposition
MeSH Terms: conditions — Psychotic Disorders; Substance-Related Disorders; Schizophrenia; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Case: Ketamine user with psychotic disorders
  Interventions: Diagnostic Test: genome testing
- Control Group 1: Ketamine user without psychotic disorders
  Interventions: Diagnostic Test: genome testing
- Control Group 2: Non-ketamine-using drug user with psychotic disorders
  Interventions: Diagnostic Test: genome testing
- Control Group 3: Non-ketamine-using drug user without psychotic disorders ( identified from register-based medical record system)

INTERVENTIONS:
Diagnostic Test: genome testing — blood sampling via venipuncture
  Groups: Case; Control Group 1; Control Group 2

SUMMARY:
Evidence suggests that repeated or chronic ketamine use, as compared to acute ketamine users, posed a higher clinical risk of developing psychotic disorders, potentially related to the underlying chronic N-methyl-D-aspartate receptor (NMDAR) dysfunction, and a higher risk of suffering from schizophrenia particularly in those genetically susceptible, or genetically predisposed ketamine abusers. With ketamine infusion rises as a emerging hope as an acute treatment for depression and suicidality under the shadow of unknown longer term psychotomimetic effects peculiarly amongst repeated or chronic use, the current case-control study aims to investigate: a) if repeated or chronic ketamine use is associated with an increased risk of psychosis by comparing those ketamine abusers with and without psychosis, and to those non-ketamine-using drug abusers with psychosis; and b) if genetic predisposition from single nucleotide polymorphisms are associated with risk of psychosis in ketamine abusers.

ELIGIBILITY:
Inclusion Criteria:

* Age: 12 - 65 years old
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Self-reported to have psychoactive substance use continuously for ≥3 month
* At least one positive urine toxicology result showing the reported psychoactive substance being used

Exclusion Criteria:

* Age <12 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed to have Intellectual Disabilities (DSM-5) or Mental Retardation (ICD-10, F70-73)
* Had been diagnosed to have primary psychosis prior to the use of any psychoactive substances, including alcohol
* Had been diagnosed to have "bipolar and related disorder" prior to the use of any psychoactive substances, including alcohol
* Had been diagnosed to have "major depressive disorder with psychotic features" prior to the use of any psychoactive substances, including alcohol
* Had been diagnosed to have "psychotic disorder due to another medical condition" (DMS-5)
* Self-reported to have abstained from any psychoactive substance use continuously for ≥12 months AND with negative urine toxicology result at the time of recruitment/ intake at the psychiatric services as recorded on case notes

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ketamine abuser and non-ketamine-using drug abusers
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
relative risk of ketamine users compared to non-ketamine using drug user to develop psychosis | During the 2 year study period
  relative risk of ketamine users compared to non-ketamine using drug user to develop psychosis

SECONDARY OUTCOMES:
Gene association to development of psychcosis | During the 2 year study period
  The single nucleotide polymorphism of 4 genes associated with N-methyl-D-aspartate and dopamine receptors being associated with the development of psychosis in ketamine abuser

CONTACTS AND LOCATIONS:
Overall Officials: albert KK Chung, MBBS(HK), Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Western Psychiatric Centre, Hong Kong